CLINICAL TRIAL: NCT05164848
Title: A Multicenter, Open-label, Phase Ib Study to Evaluate the Safety and Efficacy of JMT101 Combined With Afatinib in Patients With Advanced Esophageal Squamous Cell Carcinoma Who Have Failed Standard Therapy
Brief Title: JMT101 Combined With Afatinib in Patients With Advanced Esophageal Squamous Cell Carcinoma After Standard Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-CSP-004
Record Dates: First submitted 2021-11-03; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Squamous Carcinoma
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): JMT101 combined with two dose levels of afatinib will be tested according to the "3 + 3" dose-escalation design. The dose-limiting toxicity (DLT) will be assessed from the first administration to the end of the first cycle (28 days).
  Interventions: Drug: JMT101; Drug: Afatinib
- Dose Expansion Cohort (Experimental): Once the safe and effective dose has been determined, an expansion cohort will be recruited to further evaluate the efficacy and safety of the selected dose.
  Interventions: Drug: JMT101; Drug: Afatinib

INTERVENTIONS:
Drug: JMT101 — JMT101 will be administered intravenously at 6 mg/kg every 2 weeks (q2w) in each 28-week cycle.
Drug: Afatinib — Afatinib will be administered orally at 30 mg or 40 mg per day (qd) in each 28-week cycle.

SUMMARY:
This study is a multi-center, open-label, phase Ib study to evaluate the safety, tolerability and efficacy of JMT101 combined with afatinib in patients with advanced esophageal squamous cell carcinoma who have failed standard treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalated phase Ib study aimed to evaluate the safety, tolerability, and efficacy of JMT101 combined with afatinib in patients with advanced esophageal squamous cell carcinoma who have failed standard treatment. This study consists of two stages: dose-escalation stage and dose expansion stage. The dose-escalation stage will be conducted to determine the maximum tolerated dose (MTD) of JMT101 combined with afatinib in patients with advanced esophageal squamous cell carcinoma based on a 3+3 design. JMT101 will be given by intravenous infusion at 6 mg/kg (q2w) of each 28-week cycle. Afatinib will be sequentially administered at 30 mg and 40 mg (qd) of each 28-week cycle. One dose cohort which is verified to be well-tolerated and safe in dose-escalation stage will be selected for dose-expansion to further explore the safety, pharmacokinetic and efficacy of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or above, without gender limitation;
2. Histological or cytologically confirmed esophageal squamous cell carcinoma;
3. Patients with metastatic disease or locally advanced disease (UICC or AJCC 8th Edition) unsuitable for radical surgery or radiotherapy; with direct invasion of adjacent organs (such as aorta or trachea) (T4b) should be closely assessed for the risk of bleeding before enrollment;
4. Patients who have failed first-line or above treatments. The treatment failure is defined as disease progression or intolerable toxicity during or after the last dose of systemic standard chemotherapy, and recurrence or metastasis during treatment or within 6 months of discontinuation of radical therapy including radical concurrent chemoradiotherapy and neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy);
5. At least 1 measurable lesion according to RECIST 1.1 at baseline; if there is only one measurable lesion at baseline, the area must have not had prior radiotherapy or there must be evidence of apparent progression after radiotherapy;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
7. Life expectancy exceeds 3 months;
8. The function of major organs and bone marrow meet the following criteria within 7 days before treatment (No blood transfusion, erythropoietin (EPO), granulocyte colony stimulating factor (G-CSF), granulocyte-macrophage colony stimulating factor (GM-CSF), or other support therapy within 7 days prior to administration of the study drug):

   Blood routine: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥80×10^9/L, hemoglobin ≥80 g/L; Kidney function test: Serum creatinine ≤1.5×upper limit of normal (ULN); Liver function tests: total bilirubin ≤1.5×ULN (≤3×ULN for patients with liver metastasis), aspartate aminotransferase ( AST) and alanine aminotransferase (ALT ) ≤3×ULN ( ≤5×ULN for patients with liver metastasis); Blood coagulation: International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
9. The fertile women should have a negative blood pregnancy test within 7 days before enrollment; fertile men or women must agree to use effective contraceptive methods during the whole trial period and six months after the last administration;
10. Patients fully understand and voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

1. Previously treated with EGFR antibody;
2. Patients whose tumor has invaded important blood vessels or is much more likely to invade important blood vessels and cause fatal hemorrhage during the study according to the investigator's judgement; patients who have hemorrhage in the lung or other parts, have a bleeding tendency, or are receiving thrombolytic or anticoagulant therapy;
3. Anti-tumor therapy such as chemotherapy, biological therapy, targeted therapy, immunotherapy, etc. within 4 weeks before the first administration of the study drug; oral small molecule targeting drugs within 2 weeks of the first dose or within the 5 half-life of known drugs (whichever is longer); radiotherapy within 2 weeks before the first administration of the study drug;
4. Received other investigational product within 4 weeks before the first administration of the study drug;
5. Received major organ surgery (excluding needle biopsy) or suffered significant trauma within 4 weeks before the first administration of the study drug;
6. Received strong inducers and strong inhibitors of P-gp within 2 weeks before the first administration of the study drug;
7. Uncontrolled cancer pain; not at a stable dose of anesthetic analgesics at the time of enrollment.
8. Adverse reactions of previous anti-tumor treatments have not yet recovered to ≤ grade 1 according to CTCAE 5.0 (except for the toxicity without safety risk judged by investigator, such as alopecia);
9. Central nervous system metastasis or meningeal metastasis;
10. History of autoimmune disease or immunodeficiency disease including human immunodeficiency virus antibody (HIV-Ab) positive, or suffering from other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
11. Active hepatitis B, active hepatitis C, or positive for treponema pallidum antibodies;
12. History of severe cardiovascular disease;
13. History of other malignancies within 5 years before the first administration of the study drug, except: malignant lesions that have been treated with therapeutic measures and no known active lesions within 5 or more years before enrolment, and are judged by the treating physician to be at low risk of recurrence; adequately treated non-melanoma skin cancer and cervical cancer in situ without evidence of progression; or prostatic intraepithelial neoplasia without evidence of recurrence of prostate cancer.
14. Patients with any severe or uncontrollable disease are unsuitable to participate in this clinical trial according to the investigator's judgement;
15. Known hypersensitivity or intolerance to any component of the study drug or its excipients;
16. Past or present interstitial pneumonia/pulmonary disease;
17. Pregnant or lactating women;
18. Other situations that may increase the risks related to the study drug or affect compliance of the trial compliance are not suitable for the trial as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-25 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events，afety and Tolerability | Throughout the study period, with an average of 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).
Duration of response (DOR) | Up to approximately 2 years
  Measure of time from first response to disease progression or death
Disease control rate (DCR) | Up to approximately 2 years
  Percentage of patients who achieve partial response (PR) or complete response (CR) or stable disease (SD) based on Response Evaluation Criteria In Solid Tumors (RECIST)
Progression free survival (PFS) | Up to approximately 2 years
  Measure of time from study treatment to disease progression or death
Overall survival (OS) | Up to approximately 2 years
  Measure of time from study treatment to patient's death or lost to follow-up
Pharmacokinetic profile of JMT101 (AUC0-t) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  area under the plasma concentration versus time curve
Pharmacokinetic profile of JMT101 (Cmax) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  Peak plasma concentration
Pharmacokinetic profile of JMT101 (Tmax) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  Time for peak concentration
Pharmacokinetic profile of JMT101 ( t½) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  half life of JMT101
The incidence of anti-drug antibody (ADA) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  anti-drug antibody which can result in treatment failure by blocking the pharmacological function of the drug.
The incidence of neutralizing antibody (Nab) | Pre-dose and multiple timepoints up to 30 days after the lase dose
  neutralizing anti-drug antibody which can result in treatment failure by blocking the pharmacological function of the drug.

OTHER OUTCOMES:
The correlation of biomarkers with efficacy | Up to approximately 2 years
  The biomarkers include PIK3CA, PTEN, KRAS, BRAF, CDH1, EGFR status detected by immunohistochemical (IHC) and fluorescence in-situ hybridization (FISH).

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Anhui Provincial Hospital, Hefei, Hefei
  - Henan Cancer Hospital, Henan, Henan
  - Xinxiang Central Hospital of Henan Province, Xingxiang, Xingxiang